CLINICAL TRIAL: NCT01814319
Title: Initial Study on the Use of Probenecid as a Positive Inotrope for the Treatment of Systolic Heart Failure in Stable NYHA Class II to IV Patients
Brief Title: Repurposing Probenecid as a Positive Inotrope for the Treatment of Heart Failure
Acronym: ReProsperHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jack Rubinstein, Asst Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Re-Prosper HF
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Systolic Heart Failure
Keywords: heart failure; ejection fraction equal or less than 40%
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probenecid (Experimental): Probenecid 1 gr oral twice daily or placebo will be given to the subject for 1 week (randomly assigned). A subsequent 1 week washout period will occur followed by the alternate therapy.
  Interventions: Drug: Probenecid 1 gr oral twice daily
- placebo (Placebo Comparator): Probenecid 1 gr oral twice daily or placebo will be given to the subject for 1 week (randomly assigned). A subsequent 1 week washout period will occur followed by the alternate (placebo) therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probenecid 1 gr oral twice daily — Probenecid 1 gram oral twice daily
  Arms: Probenecid
Drug: Placebo — Matching placebo oral twice daily
  Arms: placebo

SUMMARY:
Probenecid is an FDA approved drug for the treatment gout and hyperuricemia. It has been used safely in humans for decades for this and other indications. The investigators have recently discovered that this drug can also stimulate other receptors in the heart and therefore improve its function. The hypothesis of this study is that probenecid can be used to improve the function of the heart and therefore the symptoms in patients with heart failure.

DETAILED DESCRIPTION:
The investigators will test the hypothesis that oral administration of probenecid results in improved symptomatology and heart function in patients with systolic heart failure. There will be three cohorts.

Cohort 1 will enroll up to 50 subjects in a double-blinded, randomized, placebo-control, cross-over study with each patient serving as his or her own control. The subjects will have stable HF, an ejection fraction of less than or equal to 40% and NYHA II to IV symptoms. Each subject will undergo 1 week of investigational product (IP), consisting of oral probenecid therapy 1 gram twice a day or placebo with weekly follow.

The subjects will undergo EKGs, laboratory analysis, physical exams; dyspnea and quality of life questionnaires and a 6 minute walk test (MWT) at baseline. There will be 2 optional sub-studies one for echocardiographic data and the other biomarkers.

Cohort 2 will enroll up to 50 subjects in a double-blinded, randomized, placebo-control study and will include patients admitted to the hospital with acute decompensated HF. Each subject will also receive Investigational product consisting of either 1 gram orally twice daily of probenecid or placebo during their hospitalization. They will have daily follow-up with EKG and appropriate laboratory work. In addition to the EKG, laboratory analysis, physical exams, dyspnea and quality of life questionnaires and 6 MWT data will be collected; additional data such as length of hospital stay, biomarkers, use of inotropic therapy and diuretics, and rate of diuresis will also be collected.

Cohort 3 will enroll up to 50 healthy subjects in a double-blinded, randomized, placebo-control study. Each subject will also receive Investigational product consisting of either 2 grams orally of probenecid or placebo. During a 6 hour course subjects will have laboratory analysis, physical exam, telemetry, EKG and echocardiographic studies performed as measures of both safety and effect of the compound.

ELIGIBILITY:
Inclusion Criteria

1. 18 years of age or older
2. EF < 40% via echocardiogram within the past 12 months
3. Stable dose of heart failure medications for > past 1 month
4. NYHA class II - IV

Exclusion Criteria

1. Pregnant or lactating female
2. Receiving IV inotrope
3. History of significant non-compliance
4. Unwilling to adhere to the protocol
5. Systemic systolic BP less than 90 mmHg at screening visit
6. History of allergy to probenecid
7. History of gout
8. History of renal calculi
9. Recent unstable coronary artery syndromes (USA, admission to hospital for AMI, revascularization procedure, or acute decompensated HF requiring hospitalization) within the past 3 months.
10. Implant of CRT device within the past 3 months
11. TIA, CVA or major surgery within the past 3 months
12. Valvular heart disease (more than moderate stenosis or insufficiency)
13. HOCM, myocarditis, constrictive pericarditis, congenital heart disease, 14 Active chemotherapy, significant malignancy or uncontrolled metabolic disease (untreated hyper or hypothyroidism, Cushing's disease etc.)What about uncontrolled DM?? HgA1C > etc

15. Elevated liver enzymes (> 3 times ULN), 16. Current atrial fibrillation or frequent PVCs (should we define this now) 17. End stage renal disease (dialysis dependent) or worsening renal insufficiency should define now.

18. History of gastric ulcerations, significant gastroesophageal reflux. 19. Other condition that in the opinion of the investigator, would make the subject a poor candidate for the study.

20. Co-administration of any medication that in the opinion of the investigator places the subject at increased risks due to potential adverse drug interactions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 1 week
  Measure for changes in the distance that the patient can walk over 6 minutes.
shortness of breath | 1 week
  Measure objectively if there are changes in perceived shortness of breath using a standardized scale

SECONDARY OUTCOMES:
Ejection fraction | 1 week
  We will measure via echocardiography the systolic function of the heart
beta naturietic peptide | 1 week
  We will measure for changes in the beta natuiretic peptide as a marker of cardiac function and dilatation.
serum electrolytes | 1 week
  We will measure several important electrolytes such as Na, K and Ca.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Robbins N, Gilbert M, Kumar M, McNamara JW, Daly P, Koch SE, Conway G, Effat M, Woo JG, Sadayappan S, Rubinstein J. Probenecid Improves Cardiac Function in Patients With Heart Failure With Reduced Ejection Fraction In Vivo and Cardiomyocyte Calcium Sensitivity In Vitro. J Am Heart Assoc. 2018 Jan 13;7(2):e007148. doi: 10.1161/JAHA.117.007148. PMID 29331959